CLINICAL TRIAL: NCT05127564
Title: An Open-Label, Parallel-Group, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Diroximel Fumarate (BIIB098) in Chinese and Caucasian Adult Healthy Participants
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Diroximel Fumarate (DRF) in Chinese and Caucasian Adult Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 272HV111
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — diroximel fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DRF: Chinese Participants (Experimental): Chinese participants will receive DRF Dose 1, oral capsules, twice daily (BID), from Day 1 to Day 4 and DRF Dose 1, oral capsules, once daily (QD), on Day 5.
  Interventions: Drug: Diroximel fumarate
- DRF: Caucasian Participants (Experimental): Caucasian participants will receive DRF Dose 1, oral capsules, BID, from Day 1 to Day 4 and DRF Dose 1, oral capsules, QD, on Day 5.
  Interventions: Drug: Diroximel fumarate

INTERVENTIONS:
Drug: Diroximel fumarate — Administered as specified in the treatment arm
  Other Names: Vumerity; BIIB098

SUMMARY:
The primary objective is to evaluate the primary pharmacokinetic (PK) parameters of DRF active metabolite monomethyl fumarate (MMF) following multiple doses of DRF in Chinese and Caucasian adult healthy participants. The secondary objectives are to evaluate the secondary PK parameters of DRF active metabolite MMF following multiple doses of DRF in Chinese and Caucasian adult healthy participants, to evaluate the PK of DRF inactive major metabolite 2-hydroxyethyl succinimide (HES) following multiple doses of DRF in Chinese and Caucasian adult healthy participants and to evaluate the safety and tolerability of multiple oral doses of DRF in Chinese and Caucasian adult healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilograms per meter square (kg/m^2), inclusive.
* Negative polymerase chain reaction (PCR) test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at screening and Day -1.
* For Chinese participants: was born in China, and biological parents and grandparents were of Chinese origin. If living outside China for more than 5 years, must not have had a significantly modified diet since leaving China.

Key Exclusion Criteria:

* History of severe allergic or anaphylactic reactions or of any allergic reactions that, in the opinion of the investigator, are likely to be exacerbated by any component of the study treatment; or systemic hypersensitivity reactions to DRF, dimethyl fumarate (DMF), MMF, other fumaric esters, excipients in the formulation, or diagnostic agents to be administered during the study.
* Confirmed demonstration of corrected QT interval, using Fridericia's correction method, of >450 milliseconds (ms) for males and >460 ms for females.
* Has a history of gastrointestinal (GI) surgery (except appendectomy or cholecystectomy that occurred more than 6 months prior to screening), irritable bowel syndrome, inflammatory bowel disease (Crohn's disease, ulcerative colitis), or other clinically significant and active GI condition, per the investigator's discretion.
* Has experienced clinically significant acute GI symptoms in the judgment of the investigator within 30 days prior to admission.
* History or positive test result at screening for human immunodeficiency virus (HIV).
* Chronic, recurrent, or serious infection, as determined by the investigator, within 90 days prior to screening and between screening and Day -1.
* Current enrollment in any other drug, biological, device, or clinical study or treatment with an investigational drug or approved therapy for investigational use within 30 days prior to Day -1, or 5 half-lives, whichever is longer.
* Previous participation in this study or previous studies with DRF or DMF.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Monomethyl Fumarate (MMF) | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Area Under the Concentration-Time Curve within a Dosing Interval (AUCtau) of MMF | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Concentration (Tmax) of MMF | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Elimination Half-Life (t½) of MMF | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Lag Time in Absorption (Tlag) of MMF | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Apparent Total Body Clearance (CL/F) of MMF | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Apparent Volume of Distribution (Vz/F) of MMF | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Accumulation Ratio Following Multiple Dosing (Rac) of MMF | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Maximum Observed Concentration (Cmax) of 2-Hydroxyethyl Succinimide (HES) | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Area Under the Concentration-Time Curve within a Dosing Interval (AUCtau) of HES | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Time to Reach Maximum Observed Concentration (Tmax) of HES | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Elimination Half-Life (t½) of HES | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Lag Time in Absorption (Tlag) of HES | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Apparent Total Body Clearance (CL/F) of HES | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Apparent Volume of Distribution (Vz/F) of HES | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Accumulation Ratio Following Multiple Dosing (Rac) of HES | Pre-dose and at multiple timepoints post-dose on Days 1 and 5 and post-dose on Days 6, 7 and 8
Number of Participants with Adverse Events (AEs) | Day 1 to Day 10
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants with Serious Adverse Events (SAEs) | Screening to Day 10
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- Research Site, Shatin, New Territories, Hong Kong
- Research Site, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/